CLINICAL TRIAL: NCT04338048
Title: Autosomal Dominant Polycystic Kidney Disease (ADPKD) Study
Acronym: ADPKD
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-021496
Record Dates: First submitted 2020-01-02; First posted 2020-04-08 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autosomal Dominant Polycystic Kidney Disease (ADPKD) is the most common genetic cause of renal failure. For several decades, ADPKD was regarded as an adult-onset disease. In the last decade, it has become more widely appreciated that the disease course begins in childhood. However, evidence-based guidelines on how to manage and approach children diagnosed with or at-risk for of ADPKD are lacking. Overall, there is insufficient data on the clinical course during childhood. The study intends to get more information on Autosomal Dominant Polycystic Kidney Disease (ADPKD) and other hepato/renal fibrocystic diseases. Additionally, the study intends to expand web-based resources so anyone can learn about ADPKD or other hepato/renal fibrocystic diseases. Individuals diagnosed with the dominant form of a hepato/renal fibrocystic condition are invited to be in the study.

DETAILED DESCRIPTION:
This study will ask the subject's permission to see past, current, and future medical information related to the disease. Some information that is collected, would be clinic notes, lab results, and physician consult reports. The subject will be asked to sign a release of medical information form to allow the study team access to medical information.This study does not require a clinic visit to the center.

When the research study receives the information, the research study team will be able to enter the medical data into the Hepato/Renal Fibrocystic Diseases clinical database.

There will be initial data entry in the database and follow up data entries lasting for the duration of this study or until the subject chooses to not participate in the study anymore. The study team will remove the subject's name or any other identifiable health information from the received records before entering medical data into the Hepato/Renal Fibrocystic Diseases clinical database.

ELIGIBILITY:
Inclusion Criteria:

* Demonstration of ADPKD by clinical information, imaging studies, biopsy, autopsy, or genetic testing.

Exclusion Criteria:

* Patients with Autosomal Recessive Polycystic Kidney disease (ARPKD), urinary tract malformations or major congenital anomalies of other systems suggesting a diagnosis other than recessive hepato-renal fibrocystic diseases.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients eligible are individuals diagnosed with ADPKD before the age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2030-10-30 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Database registry | up to 10 years
  Our research is designed to expand the currently limited knowledge about Autosomal Dominant Polycystic Kidney Diseases (ADPKD). Our specific goal is to create a registry of clinical information about this set of diseases.
  This study has two parts, the clinical database (medical health information) and the educational part. In this study we want to build a registry with information about ADPKD to learn more about this disease. There will be an optional urine and/or blood collection.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Guay-Woodford, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (4):
- United States (4):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Mayo Clinic, Rochester, Minnesota
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: Related Info — https://adpedkd-us.org/